CLINICAL TRIAL: NCT01010672
Title: A Phase II Study of MK-8669 When Administered as Maintenance Therapy to Japanese Patients With Metastatic Bone or Soft-tissue Sarcomas
Brief Title: Phase II Study of Ridaforolimus (MK-8669) With Metastatic Bone or Soft-tissue Sarcoma Patients (MK-8669-030 AM1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-030; 2009_688; MK-8669-030 (Other: protocol number)
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ridaforolimus 40 mg (Experimental)
  Interventions: Drug: Ridaforolimus

INTERVENTIONS:
Drug: Ridaforolimus — Ridaforolimus, oral tablet, 40 mg once daily for 5 consecutive days followed by 2-day dosing holiday each week. Participants treated until discontinuation criteria, such as progressive disease or unacceptable toxicity, were met.
  Other Names: MK-8669, AP23573, deforolimus; Ridaforolimus was also known as deforolimus until May 2009

SUMMARY:
The study evaluates efficacy of Ridaforolimus when administered as maintenance therapy to patients with metastatic bone or soft-tissue sarcoma in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologic diagnosis of bone or soft-tissue sarcoma that has metastasized, and who derive benefit following chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Completed prior chemotherapy with last dose received at least 3 and up to 12 weeks prior to randomization
* Adequate organ and bone marrow function

Exclusion Criteria:

* Presence of brain or central nervous system (CNS) metastases, unless successfully treated
* Prior therapy with rapamycin or rapamycin analogs
* Ongoing toxicity associated with prior anticancer therapy
* History or current evidence of any clinically significant disease that might confound the results of the study, complicate the interpretation of the study results, interfere with the patient's participation, or pose an additional risk to the patient

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Progression free rate (PFR) at 6 months | 6 months
  Progression free rate at 6 months is defined as the proportion of participants who are a complete response (CR, disappearance of all target lesions), partial response (PR, at least a 30% decrease in the sum of the longest diameter of target lesions) or stable disease (does not qualify for PR or progressive disease) at 6 months from the date of the first study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC